CLINICAL TRIAL: NCT06729047
Title: Prophylactic Intravenous Injection of Neostigmine Plus Atropine Versus Ketorolac on Post-dural Puncture Headache in Patients Undergoing Infraumbilical Surgeries: A Randomized Clinical Trial
Brief Title: Prophylactic Intravenous Injection of Neostigmine Plus Atropine Versus Ketorolac on Post-dural Puncture Headache in Patients Undergoing Infraumbilical Surgeries
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 04-2024-200988
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Post-Dural Puncture Headache
Keywords: Neostigmine; ketorolac
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Saline Solution; Neostigmine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Placebo Comparator): patients will receive placebo (normal saline)
  Interventions: Drug: normal Saline
- Group N (Active Comparator): patients will receive neostigmine (40 μg/kg) plus atropine (20 μg/kg)
  Interventions: Drug: Neostigmine
- Group K (Active Comparator): patients will receive ketorolac (0.5 mg/kg)
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: normal Saline — patients will receive placebo (normal saline)
  Arms: Group C
Drug: Neostigmine — patients will receive neostigmine (40 μg/kg) plus atropine (20 μg/kg)
  Arms: Group N
Drug: Ketorolac — patients will receive ketorolac (0.5 mg/kg)
  Arms: Group K

SUMMARY:
Post-dural puncture headache (PDPH) or spinal (or post-spinal) headache is one of the most common side effects of spinal anesthesia, with an incidence of 6-36%. The incidence of this complication was reported to be 76-85% after accidental dural puncture in epidural anesthesia. It usually starts within several hours after spinal anesthesia, but sometimes it can be delayed for up to 2 weeks, which usually resolves within a few days

DETAILED DESCRIPTION:
The usual symptoms of PDPH other than headache are photophobia, neck stiffness, nausea and vomiting, diplopia, tinnitus, and dizziness. The headache is usually throbbing and severe, starting from the forehead and extending to the occiput, and is aggravated by standing or sitting. This is due to meningeal traction associated with cerebrospinal fluid (CSF) pressure reduction or dilation of cerebral arteries as an indirect effect of lowering CSF pressure as a result of CSF leakage from the punctured dura. Current treatments or preventive measures for PDPH other than bed rest and hydration include theophylline, sumatriptan, caffeine, etc. In resistant or severe cases, epidural blood patch (EBP) is a well-described technique used to provide relief of pain.

The co-administration of neostigmine and atropine is a common treatment for terminating the effects of non-depolarizing muscle relaxants in the setting of general anesthesia with minimal side

ELIGIBILITY:
Inclusion Criteria:

* BMI less than 35 kg/m2
* Scheduled for infraumbilical surgeries
* American Society of Anesthesiologists (ASA) physical status: I and II

Exclusion Criteria:

1. ASA physical status more than II.
2. History of allrgic response to local anaesthetics or any of the medications used in the study
3. Patients with cognitive impairment
4. pregnancy
5. Basal body temperature of more than 38°C or less than 36°C
6. BMI more than 35 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-05 (Estimated)

PRIMARY OUTCOMES:
postdural puncture headache | 1 week
  the incidence of occurrence of PDPH in patients undergoing infraumbilical surgeries under SA.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Assiut University, Assiut, Egypt,, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kamm K, Forderreuther S. [Post-dural puncture headache]. Schmerz. 2021 Apr;35(2):139-149. doi: 10.1007/s00482-021-00540-x. Epub 2021 Mar 16. German. PMID 33725180
- [Background] Ljubisavljevic S, Zidverc Trajkovic J. Postdural puncture headache leads to clinical worsening of pre-existing chronic headache. J Clin Neurosci. 2020 May;75:30-34. doi: 10.1016/j.jocn.2020.03.043. Epub 2020 Mar 26. PMID 32223975
- [Background] Ahmadzade Z, Golparvar M, Sepiani S. Evaluation of the Preventive Effects of Neostigmine Plus Atropine on Post-Dural Puncture Headache. Adv Biomed Res. 2023 May 15;12:119. doi: 10.4103/abr.abr_81_22. eCollection 2023. PMID 37434934